CLINICAL TRIAL: NCT01719861
Title: A Phase 2a Intrapatient Dose Escalation Study of Desipramine in Small Cell Lung Cancer and Other High-Grade Neuroendocrine Tumors
Brief Title: Phase 2a Desipramine in Small Cell Lung Cancer and Other High-Grade Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Joel Neal (Other)
Responsible Party: Sponsor-Investigator, Joel Neal, Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25491; VAR0087 (Other: OnCore)
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Small Cell Lung Cancer (SCLC); Neuroendocrine Tumors
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neuroendocrine Tumors | interventions — Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Desipramine HCl (Experimental): Desipramine is a tricyclic antidepressant (TCA).
  Interventions: Drug: Desipramine HCL

INTERVENTIONS:
Drug: Desipramine HCL — Desipramine is a tricyclic antidepressant (TCA). All patients will start off with a 25 mg dose by mouth nightly (QHS), increasing weekly for 6 weeks. The target dose level at 6 weeks is 450 mg (maximum dosage) or the maximum tolerated dose (MTD) for each subject.
  Other Names: Norpramin; Pertofrane; Desmethylimipramine

SUMMARY:
Intrapatient dose escalation study of desipramine in subjects with small cell lung cancer (SCLC) and other high-grade neuroendocrine tumors.

DETAILED DESCRIPTION:
Participants will start desipramine by mouth nightly (QHS) for 6 weeks, with weekly dose escalation. Starting dose will be 25 to 75 mg. The desipramine dose will be escalated until the maximum dose of 450 mg is reached or a maximum safe dose per subject is established.

Dose level may be adjusted (decreased) based on cardiac or general adverse effects. desipramine level will be tapered if the subject experience disease progression, unless physician judges immediate suspension is in the subjects best interest.

Assessments will be conducted every 28 days, and will include ECGs, physicians and blood samples.

One partial and/or complete response will be sufficient to consider a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic small-cell lung cancer
* Metastatic high-grade neuroendocrine carcinoma of any organ system (high-grade defined by Ki-67 ≥ 20% and/or ≥ 20 mitoses/10 (HPF).
* Received at least one line of prior chemotherapy treatment for metastatic disease.
* Daily chemotherapy must be completed ≥ 2 weeks prior to registration
* Weekly chemotherapy must be completed ≥ 2 weeks prior to registration
* Chemotherapy every 2 weeks must be completed ≥ 3 weeks prior to registration
* Chemotherapy every 3 weeks must be completed ≥ 4 weeks prior to registration
* ECOG Performance Status 0 to 2
* Measurable disease by RECIST 1.1 criteria
* Age at least 18 years
* Estimated life expectancy at least 3 months
* Absolute neutrophil count ≥ 1,500/ mm³
* Platelets ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 mg/dL, OR ≤ 2 X ULN if tumor involves the liver
* AST(SGOT)
* ALT(SGPT) ≤ 3 X ULN
* Creatinine ≤ 1.5 X ULN
* Creatinine clearance ≥ 45 mL/min/1.73m²) for patients with creatinine levels above institutional normal
* QT interval corrected using Fridericia's method (QTcF) < 450 msec (males) or < 470 msec (females)
* PR < 240 msec
* QRS < 100 msec
* Brain metastases must be asymptomatic and have been adequately treated with radiation finishing at least 1 week prior to initiation of study treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Clinically-significant ventricular arrhythmia including cardiac arrest
* Myocardial infarction from coronary artery disease within 3 months of study enrollment
* Implantable pacemaker or implantable cardioverter defibrillator
* NYHA Class III or greater congestive heart failure
* Other clinically-significant cardiac disorders
* Family history of long QT syndrome.
* Concomitant or expected treatment with strong inhibitors of cytochrome p450 CYP2D6, specifically including Bupropion; Fluoxetine; or Paroxetine (must be discontinued at least 2 weeks or 5-half lives prior to the initiation of desipramine, whichever is shortest, except fluoxetine which requires at least a 5-week washout period).
* Use of medications known to increase risk of torsades de pointes, including Amiodarone; Arsenic trioxide; Astemizole; Azithromycin; Bepridil; Chloroquine; Chlorpromazine; Cisapride; Citalopram; Clarithromycin; Disopyramide; Dofetilide; Domperidone; Droperidol; Erythromycin; Flecainide; Halofantrine; Haloperidol; Ibutilide; Levomethadyl; Mesoridazine; Methadone; Moxifloxacin; Pentamidine; Pimozide; Probucol; Procainamide; Quinidine; Sotalol; Sparfloxacin; Terfenadine; Thioridazine; Vandetanib
* Other anti-depressant or anti-psychotic medications including selective serotonin re-uptake inhibitors (SSRIs); other tricyclic, monoamine oxidase inhibitors (MAOIs); serotonin-norepinephrine reuptake inhibitors (SNRIs, typical or atypical anti-psychotic)
* Metoclopramide (Reglan) because of increased risk of extrapyrimidal symptoms and neuroleptic malignant syndrome
* Symptomatic orthostatic hypotension despite adequate volume resuscitation.
* Medical history of narrow angle glaucoma
* Bipolar disorder, ongoing or active within the last 5 years
* Suicidal ideation, ongoing or active within the last 5 years
* Suicide attempt, ongoing or active within the last 5 years
* Pregnancy
* Breastfeeding
* Receiving any other investigational agents
* Any other serious or unstable concomitant systemic disorder that in the opinion of the investigator is incompatible with the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel W Neal, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 participants total were to be enrolled at Stanford Medical Center between December 2012 - December 2013
Groups:
- Desipramine HCl 25 mg: Desipramine is a tricyclic antidepressant (TCA). All patients will start off with a 25 mg dose by mouth nightly (QHS), increasing weekly for 6 weeks. By the end of the 6 weeks, patients will be taking 450 mg (maximum dosage) or a tolerable dose of desipramine without serious side effects.
Period: Cycle 1
Arm/Group | Desipramine HCl 25 mg
Started | 6
Completed | 2
Not Completed | 4
Not completed — Death | 4
Period: Cycle 2
Arm/Group | Desipramine HCl 25 mg
Started | 2
Completed | 1
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Desipramine HCl: Desipramine is a tricyclic antidepressant (TCA). All patients will start off with a 25 mg dose by mouth nightly (QHS), increasing weekly for 6 weeks. By the end of the 6 weeks, patients will be taking 450 mg (maximum dosage) or a tolerable dose of desipramine without serious side effects.
Arm/Group | Desipramine HCl
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Histology [Number; unit: participants]
  Small Cell Carcinoma of Lung | 3
  Large Cell Neuroendocrine Carcinoma of Lung | 2
  Large Cell Neuroendocrine Carcinoma of Pancreas | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) was assessed as the number of patients who achieve either a partial (PR) or complete response (CR) measured by CT scans and Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria, divided by the total number of patients treated on the study. CR: Disappearance of all target lesions, all non-target lesions, and no new lesion. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesion.
Time Frame: 6 weeks
Population: All patients who were enrolled and started therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Desipramine HCl 25 mg
Number analyzed (Participants) | 6
percentage of participants | 0

2. Secondary Outcome: Desipramine Maximum Dose
Description: Assessed as the median per patient maximum dose (MD) using intra-patient dose escalation, and reported as the highest dose of desipramine administered continuously for 1 week or greater.
Time Frame: Up to 6 weeks
Population: All patients who were enrolled and started therapy.
Measure: Median (Full Range); unit: mg daily
Arm/Group | Desipramine HCl
Number analyzed (Participants) | 6
mg daily | 75 [75 to 300]

3. Secondary Outcome: Median Serum Desipramine Levels During Treatment
Description: Median serum desipramine levels during treatment is reported as the median of the maximum steady state serum concentration observed in all patients.
  Therapeutic concentration of desipramine is 100 to 300 ng/mL, and toxic concentration is > 300 ng/mL.
Time Frame: Up to 6 weeks
Population: All patients who were enrolled and started therapy.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Desipramine HCl
Number analyzed (Participants) | 6
ng/mL | 132 [0 to 490]

4. Secondary Outcome: Progression-free Survival (PFS), Median
Description: Median PFS was defined as the time from randomization to disease progression (or death if the patient died before progression) calculated using the Kaplan-Meier method.
Time Frame: Up to 5 years from enrollment to radiographic progression or drug discontinuation
Population: All patients who were enrolled and started therapy.
Measure: Median (Full Range); unit: Months
Arm/Group | Desipramine HCl
Number analyzed (Participants) | 6
Months | 1.2 [0.2 to 3.3]

5. Secondary Outcome: Median Overall Survival (OS)
Description: Median overall survival was defined as time from enrollment to death from any cause calculated using the Kaplan-Meier method.
Time Frame: From start of enrollment until death, no limit
Population: All patients who were enrolled and started therapy.
Measure: Median (Full Range); unit: Months
Arm/Group | Desipramine HCl
Number analyzed (Participants) | 6
Months | 2.7 [1.3 to 5.6]

ADVERSE EVENTS:
Time Frame: Cycle 1 (28 days)
Arm/Group | Desipramine HCl 25 mg
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desipramine HCl 25 mg (N=6)
Death (Injury, poisoning and procedural complications) | 5 (5)
Rectal Obstruction (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desipramine HCl 25 mg (N=6)
Fatigue (General disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dry mouth (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders, Other - polyuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders, - nocturia (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
General disorders, Other - night sweats (General disorders) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
ALT increased (Investigations) | 1 (1)
AST increased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Rectal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Palpitation (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Gastrointestional disorders, other - Black stools (Gastrointestinal disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study had to be terminated early because patients with small cell lung cancer were not able to tolerate clinically relevant doses of desipramine, and no clinical activity was observed in the first enrolled patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No